CLINICAL TRIAL: NCT02017171
Title: PERL: A Multicenter Clinical Trial of Allopurinol to Prevent GFR Loss in T1D
Brief Title: A Multicenter Clinical Trial of Allopurinol to Prevent Kidney Function Loss in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alessandro Doria (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other); Joslin Diabetes Center (Other); University of Minnesota (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Toronto (Other); Northwestern University Feinberg School of Medicine (Other); Albert Einstein College of Medicine (Other); Steno Diabetes Center Copenhagen (Other); Washington University School of Medicine (Other); University of Washington (Other); Emory University (Other); University of Calgary (Other); University of Alberta (Other); University of Texas Southwestern Medical Center (Other); BCDiabetes.Ca (Network)
Responsible Party: Sponsor-Investigator, Alessandro Doria, Investigator, Joslin Diabetes Center
Organization: Joslin Diabetes Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DK101108; UC4DK101108-01 (NIH); NCT01575379 (obsolete NCT alias)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Nephropathies; Coronary Artery Disease
Keywords: Kidney Diseases; Diabetic Nephropathies; Diabetes Mellitus; Diabetes Complications; Uric acid; Allopurinol; Glomerular filtration rate; Coronary artery disease
MeSH Terms: conditions — Diabetic Nephropathies; Coronary Artery Disease; Kidney Diseases; Diabetes Mellitus; Diabetes Complications | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental): Oral allopurinol at a dose of 100 mg per day for 4 weeks and then at a dose ranging from 200 to 400 mg per day depending on kidney function
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Oral placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Arms: Allopurinol
Drug: Placebo — Inactive oral tablets identical in appearance to allopurinol tablets.
  Arms: Placebo

SUMMARY:
Despite improvements during the past 20 years in blood glucose and blood pressure control, diabetic kidney disease remains one of the most important causes of health problems in patients with diabetes. Novel treatments to complement blood glucose and blood pressure control are urgently needed. The goal of this study is to see whether a medication called allopurinol may help prevent loss of kidney function among people with type 1 diabetes. Allopurinol has been used for many years to decrease high blood uric acid and treat gout - a disease characterized by arthritis, especially of the foot joints. There is evidence suggesting that allopurinol might also be useful in people with diabetes who have normal or moderately impaired kidney function to decrease the risk of developing advanced kidney disease in the future. To prove this beneficial effect of allopurinol, we will be conducting an international clinical trial at eight diabetes centers, enrolling approximately 480 patients with type 1 diabetes who are at increased risk of developing kidney disease. Participants will be randomly assigned to take allopurinol or placebo (inactive pill) for three years, during which they will be followed through periodical visits. To prevent any possible bias, neither the participants nor the clinical staff knows who is taking allopurinol and who is taking the placebo. Kidney function will be measured at the beginning and at the end of the treatment period to see whether patients taking allopurinol experience a slower loss of kidney function over time as compared to those taking the inactive pill. If this trial is successful, the reduction in health problems resulting from the prevention or delay of kidney function loss due to the use of allopurinol would have a major impact on the lives of type 1 diabetic patients as well as on society at large, significantly reducing the human and financial costs associated with diabetic kidney disease. Because of the emphasis on early intervention, the proposed trial, if successful, will establish a new paradigm in treatments to slow or prevent progression towards end stage kidney disease in type 1 diabetes far beyond anything achieved to date.

DETAILED DESCRIPTION:
Despite improvements in the past 20 years in glycemic and blood pressure control and the introduction of 'renoprotective' drugs such as renin-angiotensin system blockers, the incidence of end-stage renal disease (ESRD) in type 1 diabetes (T1D) is not declining. Novel therapies to complement these interventions are urgently needed. Mounting evidence from prospective studies indicates that moderately elevated serum uric acid is a strong, independent predictor of an increased risk of chronic kidney disease and increased rates of loss of kidney function among T1D persons. To study whether uric acid lowering can reduce glomerular filtration rate (GFR) loss in T1D, we have established the PERL (Preventing Early Renal Function Loss in Diabetes) Consortium including investigators from Joslin Diabetes Center, the Universities of Minnesota, Colorado, Toronto, and Michigan, Northwestern University, Albert Einstein College of Medicine, and the Steno Diabetes Center in Denmark. With the support of NIH grant R03 DK094484, the Consortium has designed a three-year, multi-center, double-blind, placebo-controlled, randomized clinical trial with the specific aim of evaluating the efficacy of the urate-lowering drug allopurinol, as compared to placebo, in reducing kidney function loss among subjects with T1D. The trial is targeted to T1D patients with microalbuminuria or moderate macroalbuminuria or ongoing kidney function decline and serum uric acid levels ≥ 4.5 mg/dl, since these are the patients who are at very high risk of having rapid GFR decline and might benefit most from reductions in uric acid levels. Study subjects will be required to have a GFR between 40 and 99 ml/min/1.73 m2, consistent with the goal of intervening relatively early in the course of clinical DN rather than at later stages when structural changes are far advanced and a very large proportion of kidney function has already been lost. The primary endpoint of the study will be the GFR (as measured by iohexol plasma disappearance) at the end of a 2-month wash-out period after the 3-year intervention. Sample size calculations under various dropout and non-adherence scenarios suggest that 240 subjects in each treatment arm would provide at least 80% power to detect a clinically meaningful and achievable reduction in GFR decline in the allopurinol vs. the placebo group.If we demonstrate that allopurinol can halt or slow down GFR decline in T1D subjects, we will provide a safe and inexpensive intervention to prevent or delay kidney failure in T1D that can be applied at the earliest clinically detectable stages of renal injury. It is difficult to overstate how significant this finding would be, both from the perspective of public health and that of persons with diabetes.

Thirty-one of the 530 participants in this study were recruited as part of a pilot study (JDRF 17-2012-377, NCT01575379) and transferred to the main study (NCT02017171) when this was funded. Eligibility criteria for the pilot study were the same as those for the main study, with the exception of a wider estimated GFR interval at entry in the run-in period (eGFR=35-109) ml/min/1.73 m2) and the additional requirement of a measured GFR (iGFR) between 45 and 99 ml/min/1.73 m2 at the end of the run-in period. Pilot subjects joined the main study at a time point corresponding to the time elapsed from randomization in the pilot. Thus, they were exposed to the study medication for the same length of time (3 years) as participants who were directly enrolled in the main study. Outcomes measures were those of the main study, regardless of whether participants were transferred from the pilot or were directly enrolled in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with type 1 diabetes continuously treated with insulin within one year from diagnosis
* Duration of T1D ≥ 8 years
* Age 18-70 years
* History or presence of microalbuminuria or moderate macroalbuminuria, or evidence of declining kidney function regardless of history or presence of albuminuria and/or RAS Blocker treatment. Micro- or moderate macroalbuminuria will be defined as at least two out of three consecutive urinary albumin excretion rates [AERs] or albumin creatinine ratios [ACRs] taken at any time during the two years before screening or at screening in the 30-5000 mg/24 hr (20-3333 ug/min) or 30-5000 mg/g range, respectively, if not on RASB agents, or in the 18-5000 mg/24 hr (12-3333 ug/min) or 18-5000 mg/g range, respectively, if on RASB agents). Evidence of declining kidney function will be defined as an eGFR (CKD-EPI) decline ≥3.0 ml/min/1.73 m2/year, estimated from the slope derived from all the available serum creatinine measurements (including the one at screening assessment) from the previous 3 years. If at least 3 serum creatinine measures are not available in the previous 3 years, then the slope can be derived from creatinine values from the previous 5 years.
* Estimated GFR (eGFR) based on serum creatinine between 40 and 99.9 ml/min/1.73 m2 at screening. The upper and the lower limits should be decreased by 1 ml/min/1.73 m2 for each year over age 60 (with a lower limit of 35 ml/min/1.73m2) and by 10 ml/min/1.73 m2 for strict vegans.
* Serum UA (UA) ≥ 4.5 mg/dl at screening

Exclusion Criteria:

* History of gout or xanthinuria or other indications for uric acid lowering therapy such as cancer chemotherapy.
* Recurrent renal calculi.
* Use of urate-lowering agents within 2 months before screening.
* Current use of azathioprine, 6-mercaptopurine, didanosine, warfarin, tamoxifen, amoxicillin/ampicillin, or other drugs interacting with allopurinol.
* Known allergy to xanthine-oxidase inhibitors or iodine containing substances.
* HLA B*58:01 positivity (tested before randomization).
* Renal transplant.
* Non-diabetic kidney disease.
* SBP>160 or DBP >100 mmHg at screening or SBP>150 or DBP>95 mmHg at the end of the run-in period.
* Cancer treatment (excluding non-melanoma skin cancer treated by excision) within two years before screening.
* History of clinically significant hepatic disease including hepatitis B or C and/or persistently elevated serum liver enzymes at screening and/or history of HBV/HCV positivity.
* History of acquired immune deficiency syndrome or human immunodeficiency virus (HIV) infection.
* Hemoglobin concentration <11 g/dL (males), <10 g/dL (females) at screening.
* Platelet count <100,000/mm3 at screening.
* History of alcohol or drug abuse in the past 6 months.
* Blood donation in the 3 months before screening.
* Breastfeeding or pregnancy or unwillingness to be on contraception throughout the trial.
* Poor mental function or any other reason to expect patient difficulty in complying with the requirements of the study.
* Serious pre-existing medical problems other than diabetes, e.g. congestive heart failure, pulmonary insufficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Doria, MD, PhD, MPH, Principal Investigator — Joslin Diabetes Center; Michael Mauer, MD, Principal Investigator — University of Minnesota
Locations (30):
- United States (23):
  - Barbara Davis Center / University of Colorado Denver, Aurora, Colorado
  - Kaiser Permanente Colorado Institute of Health Research, Denver, Colorado
  - Emory University - Grady Memorial Hospital, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Brehm Center for Diabetes Research / University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Winthrop-University Hospital, Mineola, New York
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine / Montefiore Medical Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Gunderson Health System, La Crosse, Wisconsin
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Alberta Diabetes Institute, Edmonton, Alberta
  - BC Diabetes, Vancouver, British Columbia
  - LMC Diabetes and Endocrinology, Toronto, Ontario
  - Mount Sinai Hospital / University of Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Background] Ficociello LH, Rosolowsky ET, Niewczas MA, Maselli NJ, Weinberg JM, Aschengrau A, Eckfeldt JH, Stanton RC, Galecki AT, Doria A, Warram JH, Krolewski AS. High-normal serum uric acid increases risk of early progressive renal function loss in type 1 diabetes: results of a 6-year follow-up. Diabetes Care. 2010 Jun;33(6):1337-43. doi: 10.2337/dc10-0227. Epub 2010 Mar 23. PMID 20332356
- [Background] Hovind P, Rossing P, Tarnow L, Johnson RJ, Parving HH. Serum uric acid as a predictor for development of diabetic nephropathy in type 1 diabetes: an inception cohort study. Diabetes. 2009 Jul;58(7):1668-71. doi: 10.2337/db09-0014. Epub 2009 May 1. PMID 19411615
- [Background] Jalal DI, Rivard CJ, Johnson RJ, Maahs DM, McFann K, Rewers M, Snell-Bergeon JK. Serum uric acid levels predict the development of albuminuria over 6 years in patients with type 1 diabetes: findings from the Coronary Artery Calcification in Type 1 Diabetes study. Nephrol Dial Transplant. 2010 Jun;25(6):1865-9. doi: 10.1093/ndt/gfp740. Epub 2010 Jan 11. PMID 20064950
- [Background] Maahs DM, Caramori L, Cherney DZ, Galecki AT, Gao C, Jalal D, Perkins BA, Pop-Busui R, Rossing P, Mauer M, Doria A; PERL Consortium. Uric acid lowering to prevent kidney function loss in diabetes: the preventing early renal function loss (PERL) allopurinol study. Curr Diab Rep. 2013 Aug;13(4):550-9. doi: 10.1007/s11892-013-0381-0. PMID 23649945
- [Derived] Ang L, Gunaratnam S, Huang Y, Dillon BR, Martin CL, Burant A, Reiss J, Blakely P, Vasbinder A, Zhao L, Mizokami-Stout K, Tang Y, Feldman EL, Doria A, Spino C, Banerjee M, Hayek SS, Pop-Busui R. Inflammatory Markers and Measures of Cardiovascular Autonomic Neuropathy in Type 1 Diabetes. J Am Heart Assoc. 2025 Jan 7;14(1):e036787. doi: 10.1161/JAHA.124.036787. Epub 2024 Dec 27. PMID 39727210
- [Derived] Keum Y, Caramori ML, Cherney DZ, Crandall JP, de Boer IH, Lingvay I, McGill JB, Polsky S, Pop-Busui R, Rossing P, Sigal RJ, Mauer M, Doria A. Albuminuria and Rapid Kidney Function Decline as Selection Criteria for Kidney Clinical Trials in Type 1 Diabetes Mellitus. Clin J Am Soc Nephrol. 2025 Jan 1;20(1):62-71. doi: 10.2215/CJN.0000000000000567. Epub 2024 Nov 18. PMID 39423023
- [Derived] Doria A, Galecki AT, Spino C, Pop-Busui R, Cherney DZ, Lingvay I, Parsa A, Rossing P, Sigal RJ, Afkarian M, Aronson R, Caramori ML, Crandall JP, de Boer IH, Elliott TG, Goldfine AB, Haw JS, Hirsch IB, Karger AB, Maahs DM, McGill JB, Molitch ME, Perkins BA, Polsky S, Pragnell M, Robiner WN, Rosas SE, Senior P, Tuttle KR, Umpierrez GE, Wallia A, Weinstock RS, Wu C, Mauer M; PERL Study Group. Serum Urate Lowering with Allopurinol and Kidney Function in Type 1 Diabetes. N Engl J Med. 2020 Jun 25;382(26):2493-2503. doi: 10.1056/NEJMoa1916624. PMID 32579810
- See also: Study website — http://perl-study.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral placebo tablets (Inactive oral tablets identical in appearance to allopurinol tablets)
Period: Overall Study
Arm/Group | Allopurinol | Placebo
Started | 267 | 263
Completed | 205 | 217
Not Completed | 62 | 46
Not completed — Death | 10 | 4
Not completed — Withdrawal by Subject | 23 | 17
Not completed — Lost to Follow-up | 21 | 20
Not completed — ESKD | 6 | 2
Not completed — Miscellaneous | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Placebo | Total
Number analyzed (Participants) | 267 | 263 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (11.2) | 51.8 (10.6) | 51.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 95 | 179
  Male | 183 | 168 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 7 | 23
  Not Hispanic or Latino | 250 | 254 | 504
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 28 | 30 | 58
  White | 230 | 216 | 446
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 2 | 4 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI values were missing for two participants in the allopurinol group and three participants in the placebo group.
  kg/m^2
    number analyzed (Participants) | 265 | 260 | 525
    (all) | 29.5 (6.1) | 29.5 (5.9) | 29.5 (6.0)
Glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent] — Population: HbA1c values were missing for two participants in the Allopurinol group
  Percent
    number analyzed (Participants) | 265 | 263 | 528
    (all) | 8.2 (1.3) | 8.2 (1.3) | 8.2 (1.3)
Serum uric acid [Mean (Standard Deviation); unit: mg/dl] | 6.1 (1.5) | 6.1 (1.5) | 6.1 (1.5)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73 m^2] — Glomerular filtration rate estimated from serum creatinine with the CKD-EPI equation
  ml/min/1.73 m^2 | 75.4 (18.7) | 74.0 (19.4) | 74.7 (19.1)
Measured (iohexol-based) glomerular filtration rate (iGFR) [Mean (Standard Deviation); unit: ml/min/1.73 m^2] — Glomerular filtration rate measured by the plasma disappearance of an i.v. bolus of the contrast medium iohexol Population: Measured GFR value was missing for one participant in the placebo group
  ml/min/1.73 m^2
    number analyzed (Participants) | 267 | 262 | 529
    (all) | 68.7 (17.1) | 67.3 (16.7) | 68 (16.9)
Diabetes duration [Mean (Standard Deviation); unit: years] | 33.8 (12.2) | 35.3 (12.5) | 34.6 (12.3)
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 125.6 (14.7) | 126.3 (13.6) | 126.0 (14.2)
Diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 71.2 (10.4) | 71.3 (10.0) | 71.2 (10.2)
Urinary albumin excretion rate (AER) [Median (Inter-Quartile Range); unit: ug/min] — Population: Urinary AER values were missing for two participants in the placebo group.
  ug/min
    number analyzed (Participants) | 267 | 261 | 528
    (all) | 41.1 [7.7 to 216.0] | 43.0 [9.0 to 198.0] | 41.6 [8.5 to 207.5]
Albuminuria [Count of Participants; unit: Participants] — Based on overnight urinary albumin excretion rate (AER): normoalbuminuria: AER<20 ug/min, microalbuminuria: AER 20-199 ug/min, macroalbuminuria: AER => 200 ug/min Population: Urinary AER values were missing for two participants in the placebo group.
  Participants
    number analyzed (Participants) | 267 | 261 | 528
    Normoalbuminuria | 97 | 92 | 189
    Microalabuminuria | 97 | 106 | 203
    Macroalbuminuria | 73 | 63 | 136
Use of renin-angiotensin inhibitors [Count of Participants; unit: Participants] | 247 | 230 | 477
Smoking [Count of Participants; unit: Participants]
  Current | 27 | 31 | 58
  Past | 70 | 80 | 150
  Never | 170 | 152 | 322

OUTCOME MEASURES:

1. Primary Outcome: iGFR at the End of the Wash-out Period
Description: Glomerular filtration rate (GFR) at the end of the 2-month wash-out period following the 3-year treatment period, measured by the plasma disappearance of non-radioactive iohexol (iGFR) and adjusted for the iGFR at baseline.
Time Frame: End of the 2-month wash-out period following the 3-year treatment period (week 164)
Population: Intention-to-treat population with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73 m^2
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ml/min/1.73 m^2 | 61.2 [58.1 to 64.2] | 61.2 [58.1 to 64.2]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; p = 0.999, linear model for correlated errors — p value is not adjusted for multiple comparisons, a priori threshold for statistical significance: p<0.05; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-1.9 to 1.9] — Treatment difference = Allopurinol-Placebo

2. Secondary Outcome: eGFR at 4 Months of Treatment
Description: Glomerular filtration rate (GFR) at 4 months after randomization, estimated from serum creatinine and cystatin C and adjusted for the eGFR at baseline.
Time Frame: 4 months after randomization (week 16)
Population: Intention-to-treat population, with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73 m2
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ml/min/1.73 m2 | 70.3 [67.3 to 73.3] | 70.0 [67.1 to 72.9]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values. The confidence intervals are not adjusted for multiplicity and should not be used to infer treatment effects; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.6 to 2.2] — Treatment difference = Allopurinol - Placebo

3. Secondary Outcome: iGFR the End of Treatment Period
Description: Glomerular filtration rate (GFR) at the end of the 3-year treatment period, measured by the plasma disappearance of non-radioactive iohexol (iGFR) and adjusted for the iGFR at baseline.
Time Frame: End of the 3-yr treatment period (week 156)
Population: Intention-to-treat population, with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73 m2
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ml/min/1.73 m2 | 61.3 [58.3 to 64.3] | 61.0 [57.9 to 64.0]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.7 to 2.3] — Treatment difference = Allopurinol - Placebo

4. Secondary Outcome: iGFR Time Trajectory
Description: Glomerular filtration rate time trajectory estimated from iohexol disappearance GFR (iGFR) measurements at weeks 0, 80, 156, and 164. iGFR slopes were estimated by a linear mixed-effects model for longitudinal iGFR measures using a multiple imputation technique for missing values. Positive values denote increasing GFR over time, negative values denote declining iGFR over time.
Time Frame: Weeks 0, 80, 156, and 164 (from baseline to the end of washout period)
Population: Intention-to-treat population, with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73 m2/year
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ml/min/1.73 m2/year | -3.0 [-3.7 to -2.3] | -2.5 [-3.1 to -1.8]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.4] — Treatment difference = Allopurinol - Placebo. Confidence intervals are not adjusted for multiplicity and should not be used to infer treatment effects

5. Secondary Outcome: eGFR Time Trajectory
Description: Glomerular filtration rate time trajectory from baseline to end of the 2-month wash-out period (week 164) estimated from quarterly serum creatinine measurements (eGFR). eGFR slopes were estimated by a linear mixed-effects model for longitudinal eGFR measures using a multiple imputation technique for missing values. Positive values denote increasing eGFR over time, negative values denote declining eGFR over time.
Time Frame: Weeks 0, 4, 16, 32, 48, 64, 80, 96, 112, 128, 156, and 164 (from baseline to the end of washout period)
Population: Intention-to-treat population, with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73 m2/year
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ml/min/1.73 m2/year | -2.4 [-2.9 to -1.8] | -2.1 [-2.6 to -1.6]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.5] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Serum Creatinine Doubling or End Stage Renal Disease (ESRD)
Description: Risk of serum creatinine doubling or end stage renal disease (ESRD) in the allopurinol arm as compared to placebo. Results are expressed as the number of participants who experienced an event in each treatment group. The risk of an event in the allopurinol group as compared to the risk in the placebo group is expressed as hazard ratio (estimated by means of proportional hazard regression).
Time Frame: Up to the end of the 2-month wash-out period following the 3-year treatment period (Week 0 to Week 164)
Measure: Count of Participants; unit: Participants
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
Participants | 13 | 11
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.5 to 2.9] — Hazard ratio = Allopurinol / Placebo. Confidence intervals are not adjusted for multiplicity and should not be used to infer treatment effects

7. Secondary Outcome: AER at the End of the Wash-out Period
Description: Geometric mean of two urinary albumin excretion (AER) measurements at the end of the 2-month wash-out period following the 3-year treatment period, adjusted for the mean urinary AER at baseline. Results are expressed as least square means of the geometric means in each subject in each group.
Time Frame: End of the 2-month wash-out period following the 3-year treatment period (week 164)
Population: Intention-to-treat population, with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/min
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ug/min | 42.9 [24.7 to 74.4] | 31.7 [19.5 to 51.6]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values; Ratio (Final Values) = 1.4, 95% CI 2-sided [1.0 to 1.8] — Ratio = Allopurinol / Placebo. Confidence intervals are not adjusted for multiplicity and should not be used to infer treatment effects

8. Secondary Outcome: AER at the End of the Treatment Period
Description: Geometric mean of urinary albumin excretion rate (AER) during the last three months of the treatment period (Visits 15 and 16), adjusted for the mean urinary AER at baseline. Results are expressed as least square means of the geometric means in each subject in each group.
Time Frame: Last three months of treatment period (Weeks 142 and 156)
Population: Intention-to-treat population, with missing values being imputed
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/min
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
ug/min | 47.9 [32.5 to 70.6] | 37.4 [25.3 to 55.5]
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values; Ratio (Final Values) = 1.3, 95% CI 2-sided [1.0 to 1.6]; Ratio = Allopurinol / Placebo. Confidence intervals are not adjusted for multiplicity and should not be used to infer treatment effects

9. Secondary Outcome: Fatal or Non-fatal Cardiovascular Events
Description: Risk of cardiovascular events defined as the composite of CVD death (ICD-10 code I10 to I74.9), myocardial infarction, stroke (ischemic or hemorrhagic), coronary artery bypass grafting, or percutaneous coronary intervention in the allopurinol arm as compared to placebo.Results are expressed as the number of participants who experienced an event in each treatment group. The risk of an event in the allopurinol group as compared to the risk in the placebo group is expressed as hazard ratio (estimated by means of proportional hazard regression).
Time Frame: Up to the end of the 2-month wash-out period following the 3-year treatment period (week 0 to 164)
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 267 | 263
Participants | 15 | 9
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Superiority; For secondary outcomes, 95% confidence intervals are reported, without P values; Hazard Ratio (HR) = 1.9, 95% CI 2-sided [0.8 to 4.5] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: In each participants, adverse event data were collected from randomization to two months after the end of pharmacological treatment, or until study discontinuation for participants who did not complete the study. This corresponds to up to 164 weeks for participants who completed the study.
Description: The definition of Adverse Events and/or Serious Adverse Events correspond to that from the clinicaltrials.gov definitions
Arm/Group | Allopurinol | Placebo
All-Cause Mortality (participants affected / at risk) | 10/267 | 4/263
Serious Adverse Events (participants affected / at risk) | 93/267 | 82/263
Other Adverse Events (participants affected / at risk) | 121/267 | 119/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Allopurinol (N=267) | Placebo (N=263)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 5 (6)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Brugada syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 3 (4)
Coronary artery disease (Cardiac disorders) | 4 (4) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (2) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 2 (2) | 1 (2)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 3 (5)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 1 (2) | 1 (1)
Chest pain (General disorders) | 4 (5) | 2 (2)
Death (General disorders) | 2 (2) | 1 (1)
Oedema due to renal disease (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 5 (5)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 3 (3)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Herpes simplex meningitis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 4 (4)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 6 (8) | 4 (6)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 15 (18) | 13 (17)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (10)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2/84 (4) | 1/95 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1/84 (1) | 0/95 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/84 (1) | 0/95 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (6) | 8 (9)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/84 (0) | 1/95 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Amputation (Surgical and medical procedures) | 2 (2) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Debridement (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Penile prosthesis insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=267) | Placebo (N=263)
Influenza like illness (General disorders) | 17 (20) | 14 (14)
Bronchitis (Infections and infestations) | 10 (10) | 22 (27)
Sinusitis (Infections and infestations) | 16 (18) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 31 (47) | 30 (37)
Urinary tract infection (Infections and infestations) | 17 (33) | 21 (36)
Hypoglycaemia (Metabolism and nutrition disorders) | 26 (33) | 29 (47)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (17) | 16 (16)
Rash (Skin and subcutaneous tissue disorders) | 43 (58) | 39 (45)
Nasopharyngitis (Infections and infestations) | 18 (21) | 20 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT02017171/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02017171/SAP_001.pdf